CLINICAL TRIAL: NCT03367832
Title: South African Paediatric Surgical Outcomes Study (SAPSOS) A South African National, Multi-centre Fourteen Day Evaluation of Patient Care and Clinical Outcomes for Paediatric Patients Undergoing Surgery
Brief Title: South African Paediatric Surgical Outcomes Study (SAPSOS)
Acronym: SAPSOS
Status: Completed | Type: Observational
Sponsor: University of KwaZulu (Other)
Collaborators: South African Society of Anaesthesiologists (SASA) (Unknown); Safe Surgery South Africa (SSA) (Unknown)
Responsible Party: Sponsor
Other Study IDs: SAPSOS
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Anesthesia; Postoperative Complications; Child Mortality; Hospital Mortality; Pediatrics; Surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric surgical patients: All patients < 16 years, admitted to participating centres during the study period who undergo elective and non-elective surgery

SUMMARY:
There are few data of paediatric peri-operative morbidity and mortality in South Africa. There is little information on the burden or profile of surgical disease in the paediatric population, the level of anaesthesia or surgical care (specialist versus non-specialist) for paediatric patients, the quality of peri-operative care or contributing factors to poor outcomes. In order to understand current paediatric peri-operative morbidity and mortality in South Africa, it is important to start obtaining these data. Risk factors can be identified and changes can be in implemented accordingly to improve future outcomes.

The study will take place over fourteen-days. It is a South African national multi-centre prospective cohort study of paediatric patients (<16 years) undergoing surgery. The SAPSOS study (as was the South African Surgical Outcomes Study (SASOS) study) will be based on the methodology of the European Surgical Outcomes Study (EuSOS).

This study has important public health implications for South Africa as surgery is now recognized internationally as an essential part of public health, yet still needs to be defined as a priority in South Africa. Policy-makers and healthcare providers need evidence to plan resource allocation in a way that will improve quality and outcomes. The data from SAPSOS and SASOS, would provide a platform for government and health care providers in South Africa to appropriately allocate funding, make policy decisions and plan future peri-operative healthcare in South Africa.

DETAILED DESCRIPTION:
Methods

Fourteen-day, South African national multi-centre prospective cohort study of paediatric patients (<16 years) undergoing surgery.

Centres

The investigators aim to recruit from as many South African centres as possible. The investigators anticipate that every Medical University in South Africa will participate (University of Cape Town, University of the Free State, University of KwaZulu-Natal, University of Limpopo, University of Pretoria, University of Stellenbosch, Sefako Makgatho Health Sciences University, University of the Witwatersrand, and Walter Sisulu University), and most of the hospitals they support and serve will participate in this study.

Ethics approval

Ethics approval has been obtained from each university centre. This study is in effect a large scale clinical audit, and as such a waiver of consent has been approved by six of the eight medical school ethics committees, similar to the international precedent that was already set, as in the original EuSOS study, where consent was waived in 27 of the 28 European countries participating. Only the University of Witwatersrand and the University of the Free State require patient consent for SAPSOS.

Data collection and collation

Each individual centre will collect and record data on either an electronic or paper case record form (CRF) for every patient recruited. Paper CRFs will be stored within a locked office in each centre as they will include identifiable patient data in order to allow follow-up of clinical outcomes. Data will then be pseudo-anonymised by generation of a unique numeric code and transcribed by local investigators onto a secure, password protected internet based electronic CRF. Each patient will only be identified on the electronic CRF by their numeric code; thus the co-ordinating study team cannot trace data back to an individual patient without contact with the local team. A participant (patient) list will be used in each centre to match identifier codes in the database to individual patients in order to record clinical outcomes and supply any missing data points. Access to the data entry system will be protected by username and password delivered during the registration process for individual local investigators. All electronic data transfer between participating centres and the co-ordinating centre will be encrypted using a secure protocol (HTTPS/SSL 3.0 or better).

Where individual centres are unable to access the internet based case record form, pseudo- anonymised (coded) facsimile (fax) data transfer will be available to a secure, dedicated fax machine in the co-ordinating office. Pseudo-anonymised (coded) data may also be sent by mail to the coordinating centre if necessary.

Each centre will maintain a secure trial file including a protocol, local investigator delegation log, ethics approval documentation, the participant list, and other additional documentation such as trial definitions.

A final summary printout of included patients with major variables should be produced for each centre together with final data submission to double check for completeness and accuracy.

Dataset

A realistic data set will be fundamental to the success of the investigation, and this was confirmed in the EuSOS and SASOS studies where nearly complete data was available on patients. Following advice from the SASOS steering committee, the investigators have therefore adopted this dataset with minor changes applicable to paediatric patients. These key data points will not discourage centres from participating because of an excessive burden of data collection. The reliability of data collection will be analysed formally using K-statistics or intra-class correlation coefficients as appropriate.

Centre co-ordinators may request the addition of a limited number of data points to support the national SAPSOS data collection and for subsequent regional analyses. All additional data points must be discussed with the co-principal investigators and if necessary the steering committee.

Centre-specific data for each hospital will be collected once including: district/regional/tertiary centre, number of operating rooms, number of surgical, anaesthetic and intensive care unit (ICU) doctors, nurse ratios, number and level of critical care beds, availability of paediatric surgical wards, equipment appropriate to paediatric surgery and anaesthesia, availability of medication and blood, details about the reimbursement status of the hospital and public holidays or other local factors affecting patient throughput during the study period.

Sample size calculation

The investigators intend to recruit as many patients as possible in a fourteen day period, in order to establish a large, representative sample from all participating South African centres. Based on audit data from potential participating sites, the investigators believe that it is possible that the sample size may be close to 2,500 patients.

Perioperative mortality and morbidity is difficult to estimate due to the paucity of paediatric data from Middle Low Income Countries (MLIC). Assuming an overall complication rate following surgery of 5%, a sample size of 2,500 patients will yield 125 postoperative events. This will allow the inclusion of 10 to 15 variables in a logistic regression model for morbidity (including mortality and critical care admission). Statistical models may need to be adapted to the event rate provided by the sample recruited.

Statistical analysis

The data to be collected are all collected as part of routine clinical care. Categorical variables will be described as proportions and will be compared using chi-square tests. Continuous variables will be described as mean and standard deviation if normally distributed or median and inter-quartile range (IQR) if not normally distributed. Comparisons of continuous variables between groups will be performed using t-tests, one-way ANOVA or equivalent non parametric tests as appropriate. Univariate analysis will be performed to test factors associated with morbidity including planned and unplanned admission to critical care or in-hospital death.

Generalized linear mixed models using a logit link will be used to identify independent risk or prognostic factors for binary outcomes. These will include one-level models and hierarchical two-level models to account for the expected correlation in outcomes within hospitals. Data will first be analysed by Province, and then at the Country level, using Province as an independent variable. A stepwise approach will be used to enter new terms into the regression models. Factors will be entered into the models based on their univariate relation to outcome (p<0.05), biological plausibility and low rate of missing data.

Results will be reported as adjusted odds ratios (OR) with 95% confidence intervals. A single final analysis is planned at the end of the study.

Primary outcome measure

1. Incidence of in-hospital postoperative complications in paediatric surgical patients in South Africa.

Secondary outcome measures

1. Rate of mortality on the day of surgery for patients < 16 years undergoing surgery in South Africa.
2. The in-hospital mortality rate for patients < 16 years undergoing surgery in South Africa.
3. Rate of admission to critical care.

Organisation

The steering committee will be chaired by Alexandra Torborg (AT). The management team will be appointed by the Steering Committee. The duties of this team will include administration of all task projects, communication between project partners (including funders, steering committee members, national and local co-ordinators, data collation and management and preparation of reports for individual study sites. The Steering Committee is responsible for the scientific conduct and consistency of the project. The Steering Committee will ensure communication between the funder(s), study management team and co-ordinators as necessary.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients < 16 years, admitted to participating centres during the study period who undergo elective and non-elective surgery. This will include day case surgery and operative procedures outside operating theatres where a general anaesthetic (GA) is performed. -

Exclusion Criteria:

1. Patients undergoing radiological or other procedures not requiring general anaesthesia, or where general anaesthesia is performed but no procedure is done e.g. GA during a magnetic resonance imaging (MRI).
2. Obstetric surgical procedures. -

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Fourteen-day, South African national multi-centre prospective cohort study of paediatric patients (<16 years) undergoing surgery
Sampling Method: Non-Probability Sample
Enrollment: 2025 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days
  In-hospital postoperative complications in paediatric surgical patients in South Africa

SECONDARY OUTCOMES:
Mortality | 24 hours
  Rate of mortality on the day of surgery for patients < 16 years undergoing surgery in South Africa.
In-hospital Mortality | 30 days
  The in-hospital mortality rate for patients < 16 years undergoing surgery in South Africa
Critical Care | 30 days
  Rate of admission to critical care

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Torborg, MBChB, Principal Investigator — University of KwaZulu
Locations (1):
- University of KwaZuluNatal, Durban, KwaZuluNatal, South Africa

IPD SHARING:
Plan to Share IPD: Yes
On behalf of the Steering Committee, the Department of Anaesthetics, University of Kwazulu-Natal will act as custodian of the data. The Steering committee will retain the right to use all pooled data for scientific and other purposes. Members of the SAPSOS study group will have the right to access the pooled data for research purposes provided the research proposal has been reviewed and deemed satisfactory by the Steering Committee. The primary consideration for such decisions will be the quality and validity of any proposed analysis. Only summary data will be presented publicly and all institutions will be anonymised except in the individualised report provided to each institution at the end of the study. Individual patient data provided by participating sites remain the property of the respective institution.
Supporting Information: Study Protocol, ICF
Time Frame: Once the primary publications have been completed
Access Criteria: Full study protocol and ethics approval must be submitted to the Steering Committee who will then make a decision.

REFERENCES:
- [Background] LeBrun DG, Chackungal S, Chao TE, Knowlton LM, Linden AF, Notrica MR, Solis CV, McQueen KA. Prioritizing essential surgery and safe anesthesia for the Post-2015 Development Agenda: operative capacities of 78 district hospitals in 7 low- and middle-income countries. Surgery. 2014 Mar;155(3):365-73. doi: 10.1016/j.surg.2013.10.008. Epub 2013 Oct 11. PMID 24439745
- [Background] Bickler SW, Rode H. Surgical services for children in developing countries. Bull World Health Organ. 2002;80(10):829-35. Epub 2002 Nov 28. PMID 12471405
- [Derived] Torborg A, Cronje L, Thomas J, Meyer H, Bhettay A, Diedericks J, Cilliers C, Kluyts H, Mrara B, Kalipa M, Rodseth R, Biccard B; South African Paediatric Surgical Outcomes Study Investigators. South African Paediatric Surgical Outcomes Study: a 14-day prospective, observational cohort study of paediatric surgical patients. Br J Anaesth. 2019 Feb;122(2):224-232. doi: 10.1016/j.bja.2018.11.015. Epub 2018 Dec 19. PMID 30686308